CLINICAL TRIAL: NCT06878456
Title: Incidence and Management of Driveline Infection in Patients with CH-VAD: a Multi-centre, Observational Study
Brief Title: Incidence and Management of Driveline Infection in Patients with CH-VAD
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Wuhan Asia Heart Hospital (Other); Sichuan Provincial People's Hospital (Other); Zhejiang Provincial People's Hospital (Other); Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Shengshou Hu, Academician of Chinese Academy of Engineering, China National Center for Cardiovascular Diseases
Other Study IDs: China-NCCD
Record Dates: First submitted 2025-01-13; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Driveline Infection
Keywords: advanced heart failure; left ventricular assist device; driveline infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the incidence of the Driveline Infection of a novel full-magnetically levitated left ventricular assist device with a new design of driveline.

The main question it aims to answer is : The incidence of DLI in Chinese CH-VAD implanted advanced heart failure patients and the main risk factors.

CH-VAD has been approved in China for the treatment of patients with advanced heart failure.

DETAILED DESCRIPTION:
1. Background: Driveline infection (DLI) is a major complication of left ventricular assist devices (LVADs) and is associated with significant morbidity and mortality. The CH-VAD is a novel, fully magnetically levitated LVAD designed with an ultra-thin and highly flexible driveline, which may reduce the risk of DLI compared to traditional LVADs. Previous research has indicated that driveline design features, such as diameter and flexibility, are key risk factors for DLI. This study aims to assess the incidence, management, outcomes and risk factors of DLI in CH-VAD patients.Rationale: Understanding the incidence and management of DLI in patients receiving the CH-VAD can provide valuable insights into the effectiveness of this device in reducing infection rates. A better understanding of these factors will help refine clinical practices and inform device development to minimize infection risks.
2. Study Design

   * Design Type: Retrospective, observational, multicenter study.
   * Study Population: 181 consecutive patients who received CH-VAD implantations between June 2017 and October 2024 at 9 centers in China.
   * Primary Objective: To evaluate the incidence of DLI in CH-VAD patients.
   * Secondary Objectives: To identify factors associated with DLI, assess the management strategies, evaluate patient outcomes, and detect risk factors for DLI.
3. Study Population

   • Inclusion Criteria:
   * Patients who received CH-VAD implantations for advanced heart failure (AHF) between June 2017 and October 2024.

     • Exclusion Criteria:
   * No specific exclusion criteria.
4. Data Collection

   * Demographic and clinical characteristics from medical records, including age, sex, comorbidities, heart failure etiologies, INTERMACS profiles.
   * Surgical details, including device type, duration of support, and concomitant surgeries.
   * Infection prevention measures, including the use of prophylactic antibiotics, skin decolonization procedures, driveline fixation sutures, etc.
   * Driveline care measures, including dressing change frequency, types of disinfectants, dressing types, fixation measures, etc.
   * Incidence and management of DLI, including diagnostic methods, treatment approaches, and outcomes.
   * Information on the pathogens involved in DLI and complications such as recurrent infections, driveline revisions, and mortality.
5. Statistical Analysis

   * Descriptive statistics will be used to summarize patient demographics, DLI incidence, and outcomes.
   * Univariate and multivariate regression analyses will be conducted to identify potential risk factors for DLI.
   * Time-to-event analysis will be performed using Kaplan-Meier curves to evaluate freedom from DLI over time.
   * Statistical significance will be set at p<0.05.
6. Expected Outcomes and Significance

   * Primary Outcome: Incidence of DLI in patients with CH-VAD.
   * Secondary Outcomes: Risk factors associated with DLI, the impact of DLI on patient outcomes, and the effectiveness of different management strategies.
   * The findings from this study could provide valuable insights into the clinical management of CH-VAD patients and inform future advancements in LVAD design to minimize DLI.
7. Timeline

   * Study Period: June 2017 to October 2024 (Data collection period).
   * Data Analysis Period: November 2024 to January 2025.
   * Results Publication: Expected by March 2025.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received CH-VAD implantations for advanced heart failure between June 2017 and October 2024.

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 181 consecutive AHF patients who received CH-VAD implantation between June 2017 and October 2024 in China, with no patients excluded.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
the incidence of driveline infection in CH-VAD patients in China | Reported data includes baseline, peri-operative data and data at study completion. Outcome measurement is performed at the study completion, an average of 1.03 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Zhou X, Chen H, Zhang H, Zhang Y, Cui Y, Huang K, Hua Z, Yan Y, Zhou M, Zhao Q, Sun X, Wang C, Ge Z, Dong A, Hu S. Low Driveline Infection Rates in Patients With a Novel Fully Magnetically Levitated Ventricular Assist Device. Eur J Cardiothorac Surg. 2025 Dec 1;67(12):ezaf365. doi: 10.1093/ejcts/ezaf365. PMID 41137667